CLINICAL TRIAL: NCT04808661
Title: Randomized Comparison of Strategies for Uncomplicated Type B Aortic Intramural Hematoma: EndovaScular Versus mediCaL mAnagement of Type B Intramural heMatoma Trial
Brief Title: EndovaScular Versus mediCaL mAnagement of Uncomplicated Type B Intramural heMatoma Trial (ESCLAIM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Jiangmen Central Hospital (Other); Shenzhen People's Hospital (Other); Jieyang People's Hospital (Other); Hanyang University (Other); Henan Provincial Chest Hospital (Other); Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianfang Luo, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-Q-2021-004-03
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Intramural Hematoma
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Thoracic endovascular aortic repair plus optimal medical therapy
  Interventions: Procedure: Thoracic endovascular aortic repair plus optimal medical therapy
- Conservative group (Active Comparator): Optimal medical therapy
  Interventions: Drug: Optimal medical therapy

INTERVENTIONS:
Procedure: Thoracic endovascular aortic repair plus optimal medical therapy — Endovascular treatment (thoracic endovascular aortic repair) plus optimal medical therapy
  Other Names: TEVAR plus OMT
  Arms: Intervention group
Drug: Optimal medical therapy — Optimal medical therapy (strictly control of their blood pressure and heart rate)
  Other Names: OMT
  Arms: Conservative group

SUMMARY:
This trial is a multicenter, open-label and prospective randomized controlled study to compare 1-year outcomes of uncomplicated type B intramural hematoma (IMH) patients undergoing thoracic endovascular aortic repair (TEVAR) plus optimal medical therapy (OMT) with that of those undergoing OMT alone. The primary objective is to test the hypothesis that 1-year aortic-related adverse events are lower in TEVAR plus OMT group than that in OMT alone group. The secondary objective is to test the hypothesis that 1-year all-cause mortality, aortic-related mortality and re-intervention are lower in TEVAR plus OMT group than that in OMT alone group.

DETAILED DESCRIPTION:
Intervention group (TEVAR plus OMT): patients will undergo TEVAR besides strict control of blood pressure and heart rate and pain management as mentioned above. According to the preoperative imaging, the potential risk location of the aortic dissection or rupture and the extent of lesion involvement are evaluated, and the appropriate anchoring zone is selected to ensure a sufficient anchorage area of more than 15 mm. If the distance between the potential accident site and the left subclavian artery (LSA) is less than 15 mm, LSA will be covered to obtain sufficient anchoring area. LSA revascularization will be performed by chimney technique or hybrid operation, depending on the choice of the surgeon. The left femoral artery is punctured or cut, the artery sheath is inserted, and the pigtail catheter is inserted into the ascending aorta along the sheath. Next, the aortic covered stent was implanted reverse through the femoral artery under the guidance of the wire. When the stent was released, rapid pacing or intravenous antihypertensive drugs was used to ensure that the blood pressure was lower than 90 mmHg. After stent implantation, re-angiography to confirm the stent location and blood flow, which will indicate whether the operation was successful or not. After all above, the patients will be observed in the hospital for at least 3 days. Controls of the blood pressure and heart rate and relief of the symptoms will meet the discharge criteria.

Conservative group: all patients are under strict control of their blood pressure and heart rate with the guidelines-recommend drugs during hospitalization, including β receptor antagonists with or without other types of antihypertensive drugs if patients can tolerate. The target blood pressure is that systolic blood pressure fluctuates between 100-120 mmHg in the acute and sub-acute phase and blood pressure <130/80 mmHg in the chronic phase. The target heart rate should be limited to 60 bpm in the acute and sub-acute phases. Additionally, pain-releasing drugs ought to be prescribed when needed. Discharge criteria include control of the blood pressure and heart rate and relief of the symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Be confirmed as Stanford type B IMH by aorta computed tomography;
3. From onset to first clinical attach <90 days;
4. The subject or legal guardian understands the nature of the study and agrees to its;
5. provisions on a written informed consent form;
6. Availability for the appropriate follow-up visits during the follow-up period;
7. Capability to follow all study requirements.

Exclusion Criteria:

1. Persistent or recurrent pain despite full medication,;
2. Hemodynamic instability;
3. Signs of rupture (periaortic hemorrhage);
4. Depth of ULP > 10 mm;
5. Aortic diameter > 55 mm;
6. ULP around with calcification;
7. Previous history of aortic-related procedures;
8. Blunt thoracic aortic injury;
9. Iatrogenic aortic injury;
10. Inherited diseases: Turner syndrome, Marfan syndrome, Ehlers-Danlos syndrome, Loeys Dietz syndrome etc.;
11. Aortitis: Giant cell arteritis, Takayasu arteritis etc.;
12. Patients with malignant tumor whose life expectancy is less than 1 year;
13. Intolerance to endotracheal intubation and general anesthesia;
14. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of aortic-relative events | One year
  A composite of hematoma malabsorption, aorta rupture, development of aortic dissection, aortic dilatation (aortic diameter >55 mm) and ulcer-like projection >10 mm in depth.

SECONDARY OUTCOMES:
Rate of all-cause mortality | One-year
  All-cause mortality includes aortic-related and nonaortic-related mortality
Rate of aortic-related mortality | One-year
  Aortic-related death was defined as death attributable to an aortic cause during the initial admission or follow-up
Incidence of re-intervention | One-year
  TEVAR plus OMT: secondary intervention; OMT: conversion to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfang Luo, MD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- #106 Dongchuan Second Road, Yuexiu District, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohr-Kahaly S, Erbel R, Kearney P, Puth M, Meyer J. Aortic intramural hemorrhage visualized by transesophageal echocardiography: findings and prognostic implications. J Am Coll Cardiol. 1994 Mar 1;23(3):658-64. doi: 10.1016/0735-1097(94)90751-x. PMID 8113549
- [Result] Nienaber CA, von Kodolitsch Y, Petersen B, Loose R, Helmchen U, Haverich A, Spielmann RP. Intramural hemorrhage of the thoracic aorta. Diagnostic and therapeutic implications. Circulation. 1995 Sep 15;92(6):1465-72. doi: 10.1161/01.cir.92.6.1465. PMID 7664428
- [Result] Evangelista A, Dominguez R, Sebastia C, Salas A, Permanyer-Miralda G, Avegliano G, Gomez-Bosh Z, Gonzalez-Alujas T, Garcia del Castillo H, Soler-Soler J. Prognostic value of clinical and morphologic findings in short-term evolution of aortic intramural haematoma. Therapeutic implications. Eur Heart J. 2004 Jan;25(1):81-7. doi: 10.1016/j.ehj.2003.10.011. PMID 14683746
- [Result] Moral S, Cuellar H, Avegliano G, Ballesteros E, Salcedo MT, Ferreira-Gonzalez I, Garcia-Dorado D, Evangelista A. Clinical Implications of Focal Intimal Disruption in Patients With Type B Intramural Hematoma. J Am Coll Cardiol. 2017 Jan 3;69(1):28-39. doi: 10.1016/j.jacc.2016.10.045. PMID 28057247
- [Result] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Result] Nienaber CA, Kische S, Rousseau H, Eggebrecht H, Rehders TC, Kundt G, Glass A, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Fattori R, Ince H; INSTEAD-XL trial. Endovascular repair of type B aortic dissection: long-term results of the randomized investigation of stent grafts in aortic dissection trial. Circ Cardiovasc Interv. 2013 Aug;6(4):407-16. doi: 10.1161/CIRCINTERVENTIONS.113.000463. Epub 2013 Aug 6. PMID 23922146
- [Result] Fattori R, Montgomery D, Lovato L, Kische S, Di Eusanio M, Ince H, Eagle KA, Isselbacher EM, Nienaber CA. Survival after endovascular therapy in patients with type B aortic dissection: a report from the International Registry of Acute Aortic Dissection (IRAD). JACC Cardiovasc Interv. 2013 Aug;6(8):876-82. doi: 10.1016/j.jcin.2013.05.003. PMID 23968705
- [Result] Mesar T, Lin MJ, Kabir I, Dexter DJ, Rathore A, Panneton JM. Medical therapy in type B aortic intramural hematoma is associated with a high failure rate. J Vasc Surg. 2020 Apr;71(4):1088-1096. doi: 10.1016/j.jvs.2019.07.084. Epub 2020 Feb 13. PMID 32063446
- [Result] Li DL, Zhang HK, Cai YY, Jin W, Chen XD, Tian L, Li M. Acute type B aortic intramural hematoma: treatment strategy and the role of endovascular repair. J Endovasc Ther. 2010 Oct;17(5):617-21. doi: 10.1583/10-3125.1a. PMID 20939719
- [Result] Hossack M, Patel S, Gambardella I, Neequaye S, Antoniou GA, Torella F. Endovascular vs. Medical Management for Uncomplicated Acute and Sub-acute Type B Aortic Dissection: A Meta-analysis. Eur J Vasc Endovasc Surg. 2020 May;59(5):794-807. doi: 10.1016/j.ejvs.2019.08.003. Epub 2019 Dec 30. PMID 31899101
- [Result] Kitai T, Kaji S, Yamamuro A, Tani T, Kinoshita M, Ehara N, Kobori A, Kita T, Furukawa Y. Impact of new development of ulcer-like projection on clinical outcomes in patients with type B aortic dissection with closed and thrombosed false lumen. Circulation. 2010 Sep 14;122(11 Suppl):S74-80. doi: 10.1161/CIRCULATIONAHA.109.927517. PMID 20837929
- [Result] Evangelista A, Dominguez R, Sebastia C, Salas A, Permanyer-Miralda G, Avegliano G, Elorz C, Gonzalez-Alujas T, Garcia Del Castillo H, Soler-Soler J. Long-term follow-up of aortic intramural hematoma: predictors of outcome. Circulation. 2003 Aug 5;108(5):583-9. doi: 10.1161/01.CIR.0000081776.49923.5A. Epub 2003 Jul 21. PMID 12874185
- [Result] Evangelista A, Mukherjee D, Mehta RH, O'Gara PT, Fattori R, Cooper JV, Smith DE, Oh JK, Hutchison S, Sechtem U, Isselbacher EM, Nienaber CA, Pape LA, Eagle KA; International Registry of Aortic Dissection (IRAD) Investigators. Acute intramural hematoma of the aorta: a mystery in evolution. Circulation. 2005 Mar 1;111(8):1063-70. doi: 10.1161/01.CIR.0000156444.26393.80. Epub 2005 Feb 14. PMID 15710757
- [Result] Piffaretti G, Lomazzi C, Benedetto F, Pipito N, Castelli P, Trimarchi S, Dorigo W, Tozzi M. Best Medical Treatment and Selective Stent-GraftRepair for Acute Type B Aortic Intramural Hematoma. Semin Thorac Cardiovasc Surg. 2018 Autumn;30(3):279-287. doi: 10.1053/j.semtcvs.2018.02.006. Epub 2018 Feb 9. PMID 29432889
- [Result] Monnin-Bares V, Thony F, Rodiere M, Bach V, Hacini R, Blin D, Ferretti G. Endovascular stent-graft management of aortic intramural hematomas. J Vasc Interv Radiol. 2009 Jun;20(6):713-21. doi: 10.1016/j.jvir.2009.02.013. Epub 2009 Apr 23. PMID 19398351
- [Result] Felisaz A, Dufranc J, Heyndrickx M, Palcau L, Gouicem D, Berger L. Midterm results of type B intramural hematoma endovascular treatment. Ann Vasc Surg. 2015 Jul;29(5):898-904. doi: 10.1016/j.avsg.2014.12.024. Epub 2015 Feb 26. PMID 25728332
- [Result] Chen Q, Jiang D, Kuang F, Shan Z. The evolution of treatments for uncomplicated type B intramural hematoma patients. J Card Surg. 2020 Mar;35(3):580-590. doi: 10.1111/jocs.14431. Epub 2020 Jan 16. PMID 31945227
- [Result] Evangelista A, Czerny M, Nienaber C, Schepens M, Rousseau H, Cao P, Moral S, Fattori R. Interdisciplinary expert consensus on management of type B intramural haematoma and penetrating aortic ulcer. Eur J Cardiothorac Surg. 2015 Feb;47(2):209-17. doi: 10.1093/ejcts/ezu386. Epub 2014 Nov 10. PMID 25385219